CLINICAL TRIAL: NCT05248581
Title: Liver Transplantation From Living Donors For Treatment Of Non-Resectable Colorectal Carcinoma Liver Metastases: A Registry Study
Brief Title: Living Donor Liver Transplant for Unresectable Colorectal Liver Metastases
Status: Recruiting | Type: Observational
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Roberto Hernandez-Alejandro, Professor, University of Rochester
Other Study IDs: STUDY00004076
Record Dates: First submitted 2022-02-09; First posted 2022-02-21 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-06

CONDITIONS: Colorectal Cancer Metastatic
Keywords: liver transplantation; living donor; unresectable colorectal liver metastases
MeSH Terms: interventions — Liver Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — After explant of the native liver, patients will be enrolled in a biorepository with planned collection of snap frozen tissue and plasma and formalin fixed and paraffin embedded samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- All Participants: Potential subjects for this registry must have Stage IV colorectal cancer with liver metastases and be candidates for liver transplantation based on multidisciplinary discussion by the Liver transplantation team. Patients must demonstrate favorable tumor biology and no evidence of extra hepatic disease.
  Interventions: Procedure: Liver transplantation

INTERVENTIONS:
Procedure: Liver transplantation — living donor liver transplantation

SUMMARY:
The goal of this study is to create a data registry to capture clinical, pathologic, and molecular data/outcomes for patients with metastatic colorectal cancer who undergo live donor liver transplantation.

DETAILED DESCRIPTION:
The goal of this study is to create a data registry to capture clinical, pathologic, and molecular data/outcomes for patients with metastatic colorectal cancer who undergo live donor liver transplantation.

Our primary outcome of interest was the OS and recurrence-free survival (RFS) of patients who underwent LDLT at our center.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Non-amenable to curative hepatic resection as defined by FLR <30%
* Histologically confirmed adenocarcinoma of the colon or rectum
* Candidate for LDLT for colorectal liver metastasis per the University of Rochester liver transplant program

Exclusion Criteria:

* Not a candidate of the LDLT liver transplant protocol for treatment of colorectal liver metastasis.
* Unwilling to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Potential subjects for this registry must have Stage IV colorectal cancer with liver metastases and be candidates for liver transplantation based on multidisciplinary discussion by a tumor board.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2019-08-16 (Actual); Primary Completion 2027-08-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
percentage of patients with recurrence free survival | 5 years
  RFS proportions to be calculated at 1, 3, and 5 years with Kaplan Meier analysis
percentage overall survival | 5 years
  OS proportions to be calculated at 1, 3, and 5 years with Kaplan Meier analysis

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Hernandez-Alejandro, MD, Principal Investigator — University of Rochester; Matthew Byrne, MD, Study Director — University of Rochester
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided